CLINICAL TRIAL: NCT04484246
Title: Evaluation of the Incidence and Prevalence of Sarcopenia in Patients 70 Year and Older With Localized and Locally Advanced Porstate Cancer, Treated by Radiotherapy and Androgen Deprivation Therapy. a Monocentric Cohort Trial
Brief Title: Sarcopenia in Older Patient With Prostate Cancer, Prevalence and Incidence After Androgen Deprivation Therapy
Acronym: HoSAGE
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-35
Record Dates: First submitted 2020-07-06; First posted 2020-07-23 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Prevalence of sarcopenia in older patient with prostate cancer — All patients are screened for sarcopenia with the SAR-F questionnaire test score ≥4/10 suspected of sarcopenia will undergo a dual-X-ray exam to dertemine their skeletal muscle mass and the prevalence of sarcopenia before oncological treatment.

SUMMARY:
Prostate cancer is the most common cancer among men 50 years and older and mainly affets patients 75 years old.

Androgen deprivation therapy is indicatated in intermediates and high risks form of prostate cancer, in association with radiotherapy for 6 monts to 3 years. It is also indicated after surgery. Current therapies induce inhibition of sexual hormones as androgens among which testosterone. These therapies present side effects which have to be acknowledeged during the elaboration therapeutic startegies in older patients: hypogonadism induced by androgen deprivation therapy (ADT) causes loss of bone mineral density, diminution of lean body mass and increase of fat body mass.

Sarcopenia is defined by a loss of muscle strength associated to a decrease in skeletal muscle mass. In addition to aging, many factors may contribute to sarcopenia as cancer and/or ADT. This cohort study aims to evaluate risk factors associated to sarcopenia prevalence and the relationship between ADT and sarcopenia incidence, in patients 70 years or older with localized or locally advanced prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 70 years and older
* Proven localized or locally advanced prostate cancer
* Treated by radiotherapy associated to ADT
* CGA needed (screened by G8 Score ≤14)

Exclusion Criteria:

* Protected pateint under guardiaship
* Metastatic prostate cancer
* Patient refusal
* Patient cripled with severe dementia

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients 70 years or older with localized or locally advanced prostate cancer.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Prevalence of sarcopenia in older patient with prostate cancer | 36 months
  All patients are screened for sarcopenia with the SAR-F questionnaire test

SECONDARY OUTCOMES:
Evaluation of sarcopenia severity | 36 months
  The severity of the sarcopenia will be measured by the evaluation of the physical performances
Skeletal Muscular Index | 36 months
  Sarcopenia prevalence measuring Skeletal Muscular Index (SMI= Appendicular skeletal muscle mass/height²) using dual-energy X-ray absorptiometry (DXA)
Evaluation of sarcopenia severity | 36 months
  The severity of the sarcopenia will be measured by the evaluation of the muscle strength using gait speed test

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Garrido-Pradalié, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Couderc AL, Villani P, Berbis J, Nouguerede E, Rey D, Rossi D, Lechevallier E, Badinand D, Bastide C, Karsenty G, Boissier R, Amichi K, Muracciole X. HoSAGE: sarcopenia in older patient with intermediate / high-risk prostate cancer, prevalence and incidence after androgen deprivation therapy: study protocol for a cohort trial. BMC Cancer. 2022 Jan 18;22(1):78. doi: 10.1186/s12885-021-09105-8. PMID 35042460